CLINICAL TRIAL: NCT04848129
Title: What Makes Children Thin? Genetic and Behavioural Correlates of Wasting: a Pilot Study With Children Attending a Tertiary Feeding Clinic
Brief Title: Genetic Correlates of Wasting: a Pilot Study With Children Attending a Tertiary Feeding Clinic
Status: Completed | Type: Observational
Sponsor: University of Glasgow (Other)
Collaborators: University of Stirling (Other)
Responsible Party: Principal Investigator, Charlotte Wright, Professor of Community Child Health, University of Glasgow
Other Study IDs: NHSGGC290906Gen
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Undernutrition; Eating Disorders; Underweight
Keywords: Genetics; Child; Eating behaviour; Tube feeding; Avoidant Restrictive food intake disorder
MeSH Terms: conditions — Malnutrition; Feeding and Eating Disorders; Thinness; Feeding Behavior; Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Feeding clinic — These children have all attended a multidisciplinary feeding clinic with severe food refusal and were commonly receiving tube feeding or supplement drinks. The clinic helps children progress onto a normal oral diet
  Other Names: tube weaning

SUMMARY:
This is a pilot study of children attending the Glasgow feeding clinic (GFC) which looks after a range of children with severe feeding problems who commonly have low appetite and extreme thinness. The investigators want to find out if these children are more likely to carry genetic markers of thinness.

DETAILED DESCRIPTION:
Thinness occurs as a result of undereating, but it is not always clear why an individual child has not eaten enough, or how to get them to eat more. There is a need to understand the child characteristics that predispose to undereating and the how these operate, in order to design more effective treatment and prevention programmes. The Glasgow feeding clinic (GFC) looks after a range of children with severe feeding problems who commonly have low appetite and extreme thinness. The investigators want to find out if these children are more likely to carry genetic markers of thinness.

The investigators will invite up to 60 families to complete a standardised online questionnaire (ICFET) about their child's eating behaviour and collect a saliva sample from their child, sent by post. The investigators will identify how many genetic markers for thinness each carries and relate this to their ICFET appetite scores and existing growth measurements as well as their feeding history.

ELIGIBILITY:
Inclusion Criteria:

All participants currently attending Glasgow Feeding Clinic or assessed there within the last 2 years. NB current ethical application is restricted to children aged 1-7 years, but the investigators plan to apply to extend that to age 16 years.

Exclusion Criteria:

Sample not to be collected with 2 weeks of any symptoms or recent contact with Covid 19

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a heterogeneous population, united by their difficulties in eating solid food. The majority are, or have previously been, tube fed and around half have some learning disability. Thinness is very common in this group, but we will include all children, whatever their current growth pattern.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Genotype risk score | Within 1-2 months of recruitment
  This the number of risk polymorphisms present for each child ranges from 0-20. a high score suggests more thinness

SECONDARY OUTCOMES:
Eating behaviour score | At recruitment or up to 2 months before
  Measure of appetite and food refusal assessed using standard questionnaire (International Complementary Feeding Evaluation Tool (ICFET) Score from 1-5, hihger score suggests greater avidity
Body mass index | Up to two years before genetic test
  weight (kg)/Height (m) squared

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Wright, MD, Principal Investigator — University of Glasgow
Locations (1):
- New Lister building, Royal Infirmary, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The individual anonymized data would be made available on request for a collaborative genetic study
Supporting Information: Study Protocol, ICF
Time Frame: On request once initial write up is complete - after 2 years
Access Criteria: Available on request